CLINICAL TRIAL: NCT06733844
Title: Effectiveness and Acceptability Evaluation of Adolescent Nutrition CCT Pilot in Pakistan
Brief Title: Effectiveness and Acceptability of Weekly Iron Folic Acid Supplementation With Conditional Cash Transfer (WIFASCCT) Among Adolescent Girls in Four Districts of Pakistan in Low Income Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Nutrition International (Other); World Food Programme (WFP) (Unknown)
Responsible Party: Principal Investigator, Dr Sajid Bashir Soofi, Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WIFAS - CCT Study
Record Dates: First submitted 2024-11-22; First posted 2024-12-13 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Anemia
Keywords: Adolescents; anemia; weekly iron folic acid supplementations; conditional cash transfer; Pakistan
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention pilot districts (Experimental): Consisted of 4 districts from four provinces of Pakistan
  Interventions: Dietary Supplement: Weekly iron folic acid supplementations
- Control districts (No Intervention): For each intervention district within every province, a corresponding control district was selected. The control districts were identified and selected based on being the closest match to the intervention district in terms of prevalence of anemia and nutritional status (BMI) among adolescent girls as reported in the National Nutritional Survey 2018. The rate of anemia and iron folic acid intake in last pregnancy (an indicator of nutrition services being accessed) between the intervention and control districts was also comparable for the women of reproductive age (15-49 years). Comparison districts were selected for not having an ongoing WIFAS or adolescent nutrition program for adolescents.

INTERVENTIONS:
Dietary Supplement: Weekly iron folic acid supplementations — In the intervention arm, adolescent girls will receive weekly iron and folic acid supplements (WIFAS), nutrition education, and group counseling sessions. WIFAS will be delivered quarterly, with each girl consuming one supplement at the facilitation center and the remaining 12 at home, once a week. The supplements contain 60mg of iron and 2.8mg of folic acid. A quarterly cash transfer of PKR 1,000 will be given to the mother, conditional on the girl's WIFAS consumption and attendance at the quarterly education and counseling sessions. The girl will report her supplement intake at each visit and receive 13 more supplements. The intervention will last 18 months.
  Arms: Intervention pilot districts

SUMMARY:
In Pakistan, adolescent girls aged 15-19 years are particularly vulnerable to anemia and malnutrition, with over half (54.7%) being anemic. Many of these girls, especially those out of school, are often excluded from health interventions. Approximately 2.1 million adolescent girls (9%) are out of school. To address malnutrition among this group, the Government of Pakistan has prioritized adolescent girls and women under the Benazir Income Support Programme (BISP) through the Nashonuma conditional cash transfer (CCT) intervention. A new pilot program linked to the CCT is being implemented in six flood-affected districts across Pakistan. The intervention focuses on delivering nutrition interventions to adolescent daughters of Kafalat beneficiaries. This effectiveness study using a mixed-methods evaluation approach will assess the program's impact on reducing anemia, improving nutrition, and enhancing equity in access to nutrition services

DETAILED DESCRIPTION:
Introduction Adolescent girls (15-19 years) in Pakistan are among the most vulnerable to anaemia and malnutrition, with over half (54.7%) of them being anemic and living in vulnerable contexts. Among these adolescent girls, particularly those who are out of school, are often being left out by many health interventions in the country. Additionally, a significant proportion of adolescent girls, approximately 2.1 million (9%) are out of school.

The pilot intervention focuses on delivering a package of nutrition interventions to address anaemia and nutrition in adolescent daughters of Kafalat beneficiaries. It includes weekly iron and folic acid supplementations (WIFAS), nutrition education, group counselling sessions, and the provision of Weekly Iron Folic Acid Supplementation (WIFAS). WIFAS will be delivered at quarterly visits. A girl will consume one supplement at the facilitation center and then she will be recommended to consume the remaining 12 supplements, once a week on a fixed day at home. The dose of the supplements is 60mg iron and 2.8mg folic acid and once weekly continuous supplementation is recommended. A quarterly cash transfer of PKR 1,000 will be provided to the mother of the adolescent girl and the conditionality will be based on reporting consumption of WIFAS. It will also require the attendance of adolescent girls and their mothers in the quarterly nutrition education, as well as group counselling sessions at the BISP Nashonuma facilitation centers. The girl is also expected to report on her consumption at the quarterly visit and she will be given 13 more supplements to be consumed once weekly (1st supplement will be consumed at visit). This intervention is aligned with World Health Organization (WHO) recommendations for WIFAS adolescent girls in regions where anemia prevalence among women of reproductive age exceeds 20% [3]. The intervention is being delivered by the World Food Program (WFP) on behalf of BISP at the BISP Nashonuma facilitation centers.

To evaluate the impact of this new pilot program targeting adolescent girls aged 15-19 years, an effectiveness study will be carried out using a mixed-methods evaluation approach, inclusive of qualitative and quantitative research components. This evaluation aims to determine the potential to reduce anemia and to improve adolescent nutrition and equity in access to improved nutrition through the BISP conditional cash transfer program.

Objectives of the study

The proposed baseline and endline evaluation aim to evaluate the impact of the adolescent nutrition interventions and the conditional cash transfer within the CCT pilot program. The study question employing a PICO (Population, Intervention, Comparison, Outcome) framework will comprise adolescent girls of BISP Kafaalat families as 'population', WIFAS, counselling/nutrition education sessions and CCT as 'intervention' improved nutrition status, adolescent girls in BISP Kafalat households without the adolescent WIFAS, nutrition education and additional CCT as 'comparison' and hemoglobin changes, population anaemia prevalence rate (primary), and adolescent nutrition knowledge and attitudes (secondary) as 'outcome'.

The specific objectives of this evaluation study are:

* Provide Nutrition International and partners with an understanding of the effectiveness of the WIFAS, nutrition education sessions and CCT on adolescent nutrition.
* Providing an understanding of the acceptability, perspectives, experiences, and gender dynamics related to Adolescent Nutrition as a whole and the components - CCT pilot components - WIFAS, Nutrition Education and the CCT.

Complementing the stated objective, the baseline and endline evaluation study will address the following key research questions:

Primary

• What is the effectiveness of reducing anemia in adolescent girls through delivering WIFAS as part of conditional cash transfer program in 4 flood-affected districts of Pakistan?

Secondary

* Can adolescent interventions, including WIFAS (weekly iron folic supplements) and gender-responsive nutrition education be effectively delivered through conditional cash transfer programs?
* Can nutrition education be delivered to adolescents and their mothers to improve knowledge, attitudes and practices for adolescent nutrition and anaemia?
* How do nutrition education and WIFAS intervention delivered through the CCT program increase provider knowledge, awareness, and practices on adolescent nutrition?
* How does a CCT for households of adolescents influence adolescent nutrition and well-being?
* How does a CCT for households of adolescent's impact gender dynamics and decision-making and control over resources for women and adolescents?
* Which adolescents are being reached that also attend school?
* What proportion of adolescents reached through the CCT would not be reached through school-based programs?

Methodology Study design The study will employ a mixed-methods approach, employing quantitative and qualitative research methods to determine the impact, effectiveness, and effective delivery of the pilot WIFAS, nutrition education and counseling, as well as the CCT intervention.

For the quantitative assessment, repeated rounds of cross-sectional studies will be conducted at baseline and endline. The cross-sectional study design will involve random sampling of participants at each time point, both at baseline and endline, in both intervention and control districts.

For the qualitative assessment, exploratory research will guide the research design. Questions that have not been investigated to date will be explored in-depth by conducting in-depth interviews (IDIs) as well as focus group discussions (FGDs). Diversity while selecting the participants through purposive sampling will be ensured to capture a range of perspectives and experiences regarding the impact of the CCT pilot intervention and associated gender dynamics. The sample for this component will not necessarily be representative of the entire population, but internal validity will be sought.

Study sites and setting Selection of intervention districts: The intervention districts for this evaluation study will be four districts, one from each province, where the adolescent nutrition WIFAS CCT pilot program is being implemented. These districts were selected as being the most populous and feasible for study implementation, out of the 6 districts selected by the BISP and partners of the government of Pakistan as "flood-affected" districts.

The intervention districts included in the study design:

1. District Qambar Shahdadkot- Province Sindh
2. District Rajanpur - Province Punjab
3. District Lasbela - Province Balochistan
4. District Sawat - Province Khyber Pakhtunkhwa

Selection of control districts:

For each intervention district within every province, a corresponding control district was selected. The control districts were identified and selected based on being the closest match to the intervention district in terms of prevalence of anemia and nutritional status (BMI) among adolescent girls as reported in the National Nutritional Survey 2018 [6]. The rate of anemia and iron folic acid intake in last pregnancy (an indicator of nutrition services being accessed) between the intervention and control districts was also comparable for the women of reproductive age (15-49 years). Comparison districts were selected for not having an ongoing WIFAS or adolescent nutrition program for adolescents. They were also identified as "flood-affected" following the floods of August - October 2022.

Study population

The main target population for this evaluation study will be adolescent girls 15-19 years of age. The evaluation will also include the following participants:

* Mothers of the adolescent girls
* Fathers of the adolescent girls
* BISP facility providers
* Lady Health workers
* Community influencers

For the quantitative survey, the adolescent girls will be selected using the following criteria:

* From the intervention districts, adolescent girls (aged 15-19 years) who are currently living in households in the intervention communities and are recipients of: 1) Current BISP UCCT amount; 2) Additional CCT amount for having an adolescent daughter participate; 3) WIFAS for herself/adolescent daughter; and 4) Adolescent nutrition education for adolescent daughter and her mother.
* When there are multiple daughters aged 15-19 in a household, one daughter will be randomly selected using the Kish-Grid method. The Kish Grid method is a systematic approach for unbiased selection of participants in research studies. Initially, a list of eligible adolescent girls will be created and assigned a sequential number corresponding to each individual's age in ascending order. Using the Kish-Grid table with number of eligible participants and the number of households in each cluster, selection of participant will be done.
* The control group will include adolescent girls (aged 15-19 years) living in the HH in control communities and are current recipients of UCCT under Kafaalat within BISP.

Selected adolescent girls (15-19 years) will be enrolled for the Knowledge, Attitudes, and Practices (KAP) survey in the quantitative component and the collection of serum hemoglobin (Hb). Whereas a subsample of adolescent girls (50%) will be assessed for iron deficiency anemia by determining the serum ferritin, and CRP. A distinct questionnaire of knowledge attitudes and practices (KAP) will also be conducted with:

* A random subsample of 111 mothers per district and 111 fathers of the selected adolescent girls in the intervention and control districts.
* All BISP facility providers affiliated with and available at the designated BISP facilitation centers in the selected intervention districts and control districts.
* All LHWs affiliated with the designated BISP facilitation centers in the selected intervention districts.

In the qualitative component, participants will be enrolled either for In-depth interviews (IDIs) and focus group discussions (FGDs) using purposive sampling in the intervention districts.

IDIs will be conducted with the following participants:

* Adolescent girls (15-19 years)
* Mothers of adolescent girls
* Fathers of adolescent girls
* BISP facility workers
* Lady health workers

FGDs will be conducted with the following participants:

• Community influencers

ELIGIBILITY:
Inclusion Criteria:

* Adolescent girls 15-19 years of age
* Currently living in households in the intervention communities
* Their mothers are current recipients of the BISP UCCT amount
* Their mothers are current recipients of Additional CCT amount for having an adolescent daughter participate
* Receiving WIFAS for herself and for her adolescent daughter
* Participate in adolescent nutrition education sessions.
* Mothers of adolescent girls
* Fathers of adolescent girls
* BISP facility providers
* Lady Health workers
* Community influencers

Exclusion Criteria:

* Adolescent girls (aged 15-19 years) who are not currently living in households in the intervention communities
* Are not recipients of the current BISP UCCT amount, and additional CCT amount for having an adolescent daughter.

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Adolescent girls
Enrollment: 2131 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Anemia prevalence rate among adolescent girls | At 18 months

SECONDARY OUTCOMES:
Effectiveness of delivery | At 18 months
  This outcome will measure whether provision of Weekly Iron Folic Acid Supplements (WIFAS) through conditional cash transfer programs along with nutrition education can be effective in reducing anemia among adolescent girl.
Knowledge, Attitudes, and Practices (KAP) to adolescent nutrition and anemia | At 18 months
  This outcome will measure the improvement in knowledge, attitudes, and practices (KAP) related to adolescent nutrition and anemia among adolescents and their mothers after nutrition education. The changes in KAP will be assessed by comparing the intervention and control groups, as well as by comparing baseline and endline findings within the intervention group.
Impact of the conditional Cash Transfer (CCT) program on Women's Empowerment | At 18 months
  This outcome will look at how the CCT program affects gender roles, especially in terms of women's and adolescents' control over decision-making and resources. It will measure how the program influences who makes important decisions in the household and how much control women and adolescents have over money and other resources.
Proportion of School-Attending and Out-of-School Adolescents Reached by the CCT Program | At 18 months
  Description: This outcome will measure the proportion of both school-attending and out-of-school adolescents reached by the Conditional Cash Transfer (CCT) program. It will identify and compare the participation rates of adolescents in both groups, assessing the program's effectiveness in reaching a broader adolescent population beyond school-based settings.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan